CLINICAL TRIAL: NCT06719778
Title: Prospective Interventional Study to Evaluate the Impact of Diet and Lifestyle Modification on the Intestinal Barrier Integrity in Crohn's Disease
Brief Title: Impact of Diet and Lifestyle Modification on the Intestinal Barrier Integrity in Crohn's Disease
Acronym: LeakyDiet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Heidelberg University (Other); German Crohn's and Colitis Association (DCCV e.V.) (Unknown)
Responsible Party: Principal Investigator, Jost Langhorst, Univ. Prof. Dr. med, Universität Duisburg-Essen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23067
Record Dates: First submitted 2024-11-26; First posted 2024-12-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Crohn's Disease
Keywords: integrative medicine; lifestyle modification; intestinal barrier; Mediterranean diet; inflammatory bowel disease; Confocal Laser Endomicroscopy; Crohn Disease; microbiome; nutrition; irritable bowel
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Application of a two-stage nutritional therapy concept (Experimental): Sequencing of the inpatient integrative medicinal lifestyle modification program applied at the clinic for internal and integrative medicine in Bamberg into a two-stage nutritional therapy concept
  Interventions: Other: Two-stage nutritional therapy concept

INTERVENTIONS:
Other: Two-stage nutritional therapy concept — 1. Stabilization phase:
     application of a mostly vegetarian Mediterranean wholefood diet and strategies from a comprehensive lifestyle modification concept.
  2. Elimination phase:
  additional omission diet avoiding the food that was identified by CLE to induce an intestinal barrier defect.

SUMMARY:
The goal of this prospective interventional study is to evaluate whether the targeted avoidance of a particular food that was diagnosed to be disruptive for the intestinal barrier during confocal laser endomicroscopy (CLE) contributes significantly to stabilizing the intestinal barrier and improving abdominal symptoms, quality of life and disease activity in Crohn's Disease patients with food-related symptoms.

The main questions the study aims to answer are:

* whether a food-induced intestinal barrier disorder in Crohn's disease patients can be detected by endoscopy using confocal laser endomicroscopy (CLE) and a causal relationship with certain foods can be established.
* whether a change in diet or a targeted elimination diet can restore the defective integrity of the intestinal barrier detected by CLE.
* to examine whether a targeted avoidance of a food that was identified by CLE to trigger intestinal barrier disruption leads to a relevant improvement in symptoms, quality of life and disease activity in patients with Crohn's disease.

Participants will undergo a two-stage nutritional therapy concept based on a two-week inpatient integrative medicinal lifestyle modification program that comprises nutritional therapy, stress management strategies, mind-body medicine, herbal medicine and exercise:

* Initially, participants learn how to employ the comprehensive lifestyle modification concept and receive nutritional training on a mostly vegetarian Mediterranean wholefood diet.
* In a first stabilization phase, lasting for 3 months, participants independently apply the taught Mediterranean diet and use strategies from the comprehensive lifestyle modification program.
* In a second elimination phase, lasting for another 3 months, participants additionally avoid the particular food that was identified by CLE to induce an intestinal barrier defect.

Crohn's disease patients will:

* initially receive a clinically indicated endoscopy with CLE and food challenge to examine whether a food-induced intestinal barrier disorder is present
* return to the clinic for an optional endoscopy with CLE and food challenge after the first (stabilization) phase as well as the second (elimination) phase
* answer questionnaires at study start as well as after the first and the second study phase to analyze their quality of life, the severity of their symptoms and their disease activity
* give samples of blood, urine, stool and bile fluid as well as intestinal biopsies during regular inpatient sampling at study start as well as after the first and the second study phase
* document their intake of food and their symptoms in an App-based diary throughout the study participation

DETAILED DESCRIPTION:
Background: Chronic inflammatory bowel diseases (IBD) are multifactorial diseases in which diet can have both a positive and a negative influence. While, on the one hand, a switch to a Mediterranean plant-based wholefood diet has been shown to improve symptoms, quality of life and disease activity through a better supply of anti-inflammatory micronutrients and fatty acids, on the other hand diet is perceived by around two thirds of IBD patients as a symptom trigger. The leaky gut hypothesis offers a possible mechanistic explanation of this correlation. It describes how microbial pathogens or their components, but also food can reach deeper cell layers of the intestine through intestinal barrier disorders ("leaky gut"). There, they trigger immune reactions contributing to or driving food intolerances, allergies and IBD. To date, the functional relationship between food-induced intestinal barrier disorders and symptoms in Crohn's disease (MC) patients has not been investigated due to a lack of technical feasibility. Confocal laser endomicroscopy (CLE) is the first technology that makes it possible to observe the intestinal barrier on site in the intestine during routine endoscopy in real time at 1000x magnification and thus to functionally check whether the application of certain foods has an effect on the intestinal barrier.

Aim: The aim of the presented prospective interventional study is to investigate in an inpatient initiated two-stage nutritional therapy concept whether the targeted avoidance of a food that was identified by CLE to disrupt the intestinal barrier, contributes significantly to the stabilization of the intestinal barrier and improvement of abdominal symptoms, quality of life and disease activity in MC patients with food-related symptoms when compared to a pure lifestyle modification including a mostly vegetarian Mediterranean wholefood diet.

Study design: For this purpose, 30 MC patients with suspected food-related symptoms are initially examined via CLE (during a routine esophagogastroduodenoscopy of the inflammation-free duodenum) to determine whether they react to the five most common food allergens wheat, yeast, milk, soy and egg white ("food challenge") with an intestinal barrier disorder. If a food-related intestinal barrier disorder is detected, a 2-stage nutritional therapy concept is applied. The 2-stage nutritional therapy concept consists of a stabilization phase (Phase 1) and an elimination phase (Phase 2). Phase 1 comprises a 3-month period during which the participants apply a mostly vegetarian Mediterranean whole-food diet and use strategies from an integrative medicinal lifestyle modification program that comprises nutritional therapy, stress management strategies, mind-body medicine, herbal medicine and exercise initially taught during detailed initial training at the clinic for internal and integrative medicine in Bamberg. Phase 2 comprises another 3-month period during which the participants particularly avoid the food that was identified by CLE to induce an intestinal barrier defect while they stay on the diet and apply the comprehensive lifestyle modification concept taught and applied during Phase 1. Throughout the study, participants document their nutrition and symptoms in a digital food and symptom diary with integrated questionnaire query via app. At the end of the first and the second phase, a CLE is used to check whether there is still a food-induced intestinal barrier disorder.

To assess the effect of the two therapy phases, clinical questionnaires are collected at the beginning and end of each phase (at week 0, W12, W24) to record IBD-specific, nutrition-related and general quality of life, symptoms, disease activity, fatigue and stress levels, as well as dietary behavior. In addition, blood, stool, urine, bile and biopsy samples are taken for examination. These serve to clarify mechanistic relationships between the intestinal barrier function, the microbiome, its metabolic products (metabolome), the systemic allergy status, the immune system and the inflammatory process (inflammation markers, immune cells and cytokines), and thus for the potential identification of diagnostic markers that can be used on an outpatient basis. The statistical comparison of the two phases is intended to examine whether the additional, targeted avoidance of foods identified by CLE as disruptive to the intestinal barrier can make a substantial contribution to stabilizing the intestinal barrier and improving abdominal symptoms, quality of life and disease activity in MC patients with food-related symptoms compared to a pure Mediterranean plant-based wholefood diet.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years
* Crohn's Disease for at least 6 months (date of initial diagnosis)
* with suspected food-induced symptoms or irritable bowel syndrome-like symptoms (fulfils IBS-Rom-IV criteria) for at least 3 months with moderate to severe symptom severity
* stable IBD-specific medication dosage for at least 3 months [such as 5-aminosalicylates (5-ASA), thiopurines or biologicals (therapeutic antibodies such as infliximab, adalimumab, vedolizumab, etc.)].
* inpatient admission to the clinic for internal and integrative medicine in Bamberg for regular treatment
* clinical indication and performance of an initial esophagogastroduodenoscopy with confocal laser endomicroscopy with detection of a food-induced intestinal barrier disorder
* signed informed consent form

Exclusion Criteria:

* severe flare of Crohn's disease
* artificial intestinal outlet
* IgE-mediated type 1 allergy to CLE-tested foods (egg white, soy, milk, yeast, wheat)
* macroscopic inflammation of the duodenum (detected via endoscopy)
* pregnancy or breastfeeding
* chronic alcohol or drug abuse
* treatment with antibiotics within one month before the start of the study
* Acute or chronic infectious, inflammatory or autoimmune intestinal diseases (such as coeliac disease, Whipples disease, lambliasis, eosinophilia, ulcerative colitis, infectious enterocolitis) or other organs (such as chronic hepatitis, autoimmune hepatitis, rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis)
* malignant diseases affecting internal organs within the last 5 years (such as colorectal cancer, stomach cancer, pancreatic cancer, liver cancer, lung cancer, breast cancer)
* severe mental disorders that impair the participant's ability to understand or follow the study protocol (e.g. uncontrolled schizophrenia, severe bipolar disorder, severe depression)
* inability to give written consent or follow study protocols
* participation in another therapeutic study within the last 30 days (except health services research)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Improvement of the integrity of the duodenal intestinal barrier analyzed by confocal laser endomicroscopy (CLE) | week 0, 12, 24
  The integrity of the intestinal barrier is tested by CLE during routine Oesophagogastroduodenoscopy. By CLE, the intestinal mucosa and the epithelial lining can be analyzed in vivo with a 1000 x magnification. An intestinal barrier defect can be detected by the leakage of a contrast agent (fluorescein) from the blood vessels through the intestinal epithelial spaces into the intestinal cavity and the shedding of epithelial cells. The impact of 5 foodstuffs (egg white, soy, milk, yeast, wheat) on the intestinal barrier is tested subsequently.
  The integrity of the intestinal barrier and the reaction to the 5 foodstuffs is tested at baseline as well as after phase 1 (at week 12) and after phase 2 (week 24) in order to identify whether a dietary change or the omission of a particular foodstuff that was identified by baseline CLE to be intestinal barrier disrupting, lead to a relevant improvement in barrier integrity.

SECONDARY OUTCOMES:
Severity of IBS symptoms by IBS-SSS (Irritable Bowel Severity scoring system) | week 0, 12, 24
  5-item questionnaire with a scale from 0 % (= not at all) to 100 % (= very severe) with a total score ranging from 0 - 500 to evaluate the severity of IBS symptoms. Use of a cut off of IBS-SSS scores to evaluate the severity of IBS: less than 175 for mild IBS, 175-300 for moderate IBS, more than 300 for severe IBS
Severity of IBD-SI (Inflammatory Bowel Disease Symptom Inventory) | week 0, 12, 24
  The IBD-SI combines items from existing clinician-rated or diary-format inventories. After factor analysis, 38 items were retained on 5 subscales: bowel symptoms, abdominal discomfort, fatigue, bowel complications and systemic complications. A total score as well as subscale scores will be calculated. Higher scores indicate more severe symptoms. Each item is scored between 0 and 4. The total score is calculated by summing the item scores together. Subscale scores are calculated by summing up the scores of particular items (bowel and systemic complications subscales) or by calculating the mean item score across the items of each of these subscales (bowel symptoms, abdominal discomfort, fatigue symptoms subscales).
Severity of HBI (Harvey-Bradshaw-Index) | week 0, 12, 24
  The disease severity of CD patients is evaluated via a validated questionnaire that is specific for Crohn's Disease (Harvey-Bradshaw-Index): The HBI was designed as a simplified version of the CDAI to enable systematic collection of clinical data on Crohn's disease and is used to assess the degree of illness in individuals with Crohn's disease.
  The index considers five, exclusively clinical parameters. A specific score is assigned for each parameter. To assess disease activity, the sum score is formed from questions on general condition, abdominal pain, number of unformed bowel movements per day, abdominal resistance and complications.
  The highest possible sum is 30 points and indicates a severe course of disease. A lower sum than 5 points indicates a clinical remission.
Disease-specific quality of life by IBD-Q (Inflammatory Bowel Disease Questionnaire) | week 0, 12, 24
  The IBD-Q is the most frequently used questionnaire for disease-specific quality of life in clinical studies on Crohn's disease. It operationalizes quality of life on 4 dimensions (emotional and social impairment as well as bowel-related and systemic symptoms), in addition to a sum score.
  Answers are recorded on a 7-point Likert scale. High values mean good, low values a reduced quality of life (1=worst score, 7=best score). The total IBD-Q scale ranges from 32 to 224. A score of ≥ 170 can be considered as normal quality of life.
Diagnosis of functional bowel disorders using Rome IV criteria | week 0, 12, 24
  Rome IV criteria were created by the Rome Foundation and are used to diagnose functional bowel disorders, including irritable bowel syndrome. They refer to symptoms (abdominal pain) that must persist over a period of at least three months and are associated with changes in bowel habits (defecation, change in frequency of stool, change in form of stool). These criteria allow a comprehensive assessment of the functional bowel status of the patients in this study.
Assessment of health-related quality of life with the Short Form 12 Health Survey (SF-12) | week 0, 12, 24
  The Short Form 12 Health Survey (SF-12) is a validated tool with 12 questions for the general assessment of the physical and mental health status of patients that is widely used in clinical studies. It is the shorter version of the SF-36 questionnaire. Two scores - one score for the physical component (PCS) and one score for the mental component (MCS) - represent the results. The SF-12 physical scale score represents general health perception, physical functioning, physical role functioning, and pain. The mental health score reflects emotional role functioning, mental well-being, negative affectivity, and social functioning. The values determined are compared with the values of the normal population with a mean of 50 and a standard deviation of 10 in the general population. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.
Assessment of the severity of the fatigue syndrome with the Multidimensional Fatigue Inventory (MFI-20) | week 0, 12, 24
  The Multidimensional Fatigue Inventory (MFI) is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity and mental fatigue. The German validated version is used. A scale from 1 to 5 is used to indicate how aptly certain statements regarding fatigue represent the participants' experiences. Higher total scores correspond with more acute levels of fatigue. Each dimension consists of four questions. The dimensional score consequently ranges from 4 to 20.
Assessment of perceived stress using the Perceived Stress Scale (PSS-10) | week 0, 12, 24
  The Perceived Stress Scale (PSS-10) is a well-established self-report scale and an international standard instrument for measuring perceived stress. The ten questions ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way on a five-point scale from 'never' to 'very often'. The PSS score is obtained by summing across all items after responses to the four positively stated items have been reversed. Higher scores indicate higher levels of perceived stress.
Assessment of anxiety and depression using the Hospital Anxiety and Depression Scale (HADS) | week 0, 12, 24
  Anxiety and depression are measured using the Hospital Anxiety and Depression Scale (HADS). The HADS was developed specifically for physically ill patients in clinical settings. The questionnaire contains 14 items: 7 on the anxiety and 7 on the depression scale. The sum values of the HADS-A (anxiety) and HADS-D (depression) scales lie in the 0-21 range, with higher values indicating a stronger manifestation of anxiety/depressiveness. The German validated version is used.
Assessment of food-related quality of life using the FR-QoL-29 questionnaire | week 0, 12, 24
  A validated questionnaire for the systematic assessment of food-related quality of life (FR-QoL) in IBD patients is used to assess psychosocial factors in connection with eating and drinking, such as enjoying food, managing restrictions, and maintaining social relationships. The FR-QoL-29, which contains 29 items, each scored on a 5-point Likert scale (1 = strongly agree; 2 = agree; 3 = neither agree nor disagree; 4 = disagree; 5 = strongly disagree), with 4 questions reversed for scoring. Scores are summed, with a total possible score ranging from 29 to 145, where higher scores reflect a greater FR-QoL.
Assessment of frequency of consumption and usual portion sizes of particular food groups using the DEGS-Food Frequency Questionnaire | week 0, 4, 8, 12, 16, 20, 24
  A food frequency questionnaire (FFQ) is used to determine the frequency of consumption and usual portion sizes of a total of 53 food groups consumed in the last four weeks. The dietary questionnaire was developed and validated for the use in the German Health Examination Survey for Adults 2008-2011 (DEGS). In this study it is used to assess whether the participants' dietary habits change throughout the study and whether they apply the diet taught during nutritional therapy at the inpatient stay at the Clinic for internal and integrative medicine in Bamberg.
Patient diary | week 0 to week 24
  Over the course of the study, the participants keep a digital diary in the form of an application on their smartphone. This application is used as a nutritional diary for the documentation of the participants' daily intake of food and the contained ingredients as well as a symptom diary for the documentation of signs of disease, stool consistency and overall well-being. The nutritional diary is used to assess whether the participants' dietary habits change throughout the study, whether they avoid the particular food that led to a disruption of the intestinal barrier during CLE and whether they apply the diet taught during nutritional therapy at the inpatient stay at the Clinic for internal and integrative medicine in Bamberg. The symptom diary is used to evaluate whether food-related symptoms can be reduced in the course of the study and this can be correlated with a stabilization of the intestinal barrier (determined during confocal laser endomicroscopy).
Oesophagogastroduodenoscopy (OGD) with confocal laser endomicroscopy (CLE) | week 0, 12, 24
  At week 0, participants undergo an OGD with CLE when clinically indicated as part of their inpatient care. Thereby, the inflammatory status and the intestinal barrier is routinely analyzed. Participants return for a voluntary OGD with CLE at week 12 and week 24. The data collected from the initial examination at week 0 is compared to the data from week 12 and week 24. Confocal laser endomicroscopy (CLE, Cellvizio System from Mauna Kea Technology) is the first technology that enables live characterization of the intestinal mucosa and barrier integrity at the cellular level during endoscopy at up to 1000x magnification, allowing local intestinal barrier disorders to be identified and targeted biopsies to be taken. This combined examination of endoscopy and CLE thus enables a comprehensive assessment of the intestinal mucosa on a macroscopic, microscopic and functional level in real time.
Histopathological analysis of duodenal biopsies | week 0, 12, 24
  Intestinal biopsies, which are routinely taken during oesophagogastroduodenoscopy, are processed for histopathological analysis of the mucosal and epithelial structure as well as of the immune cell compartment (H&E staining).
Immunohistochemical analysis of duodenal biopsies | week 0, 12, 24
  Intestinal biopsies, which are routinely taken during oesophagogastroduodenoscopy, are stained using immunohistochemistry and examined for the expression of specific marker proteins. For example, the intestinal barrier will be examined by immunohistochemical analysis of the tight junction marker proteins occludin and claudin-2 or the migration of specific immune cells such as T-lymphocytes using CD3 staining.
Gene expression analysis of duodenal biopsies | week 0, 12, 24
  Intestinal biopsies taken in addition to those routinely taken during oesophagogastroduodenoscopy are used for transcriptional analysis by q-PCR to study the gene expression of particular immune cell or inflammatory marker proteins as well as tight junction proteins.
Evaluation of the systemic inflammatory status by analysis of serum-cytokine concentrations | week 0, 12, 24
  To evaluate the systemic inflammatory status, the level of various cytokines such as IL-1β, IL-6, IL-8, IL-10, TNF, IFN-γ, IL-17or IL-4 is analyzed in the serum.
Evaluation of the complete blood count | week 0, 12, 24
  A complete blood count is made. It provides information about the number and type of immune cells. In combination with the general inflammatory markers C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR), the complete blood count allows conclusions about the presence and extent of systemic inflammation as well as the disease activity.
C-reactive protein (CRP) in the blood | week 0, 12, 24
  The concentration of the inflammation marker CRP is measured in the blood.
Erythrocyte Sedimentation Rate (ESR) | week 0, 12, 24
  Determination of the ESR of the blood.
IgE and IgG/IgG4 screening of antibodies against typical food allergens in the serum | week 0
  The serum concentrations of a total of 22 food allergen-specific IgE and IgG/IgG4 antibodies are measured in order to examine a possible connection to the food-induced intestinal barrier disorders.
anti-ASCA (anti-Saccharomyces-cerevisiae antibodies) | week 0
  Anti-ASCA (anti-Saccharomyces cerevisiae antibodies) are measured in serum samples. Anti-ASCA are analyzed to help diagnose and differentiate the inflammatory bowel disease, as they are common in patients with Crohn's disease but less common in ulcerative colitis or other bowel conditions. The measurement will be used to specify the patient collective and to investigate the connection to the intestinal barrier disorder induced by baker's yeast (Saccharomyces cerevisiae).
Lymphocyte-transformation test (LTT) | week 0
  T-lymphocytes are isolated from blood samples and are stimulated with 20 different staple foods in order to detect T-lymphocytes that react to one of the tested antigens specifically (Lymphocyte-transformation test (LTT)).
  These functional food stimulation assays with immune cells will be performed to investigate potential links between the occurrence of food-induced intestinal barrier dysfunction and the hitherto unknown pathophysiology.
Flow CAST | week 0
  Basophilic granulocytes are key cells in the allergic immune response. Therefore, the activation of basophils is analyzed in blood samples in order to analyze whether these cells play a role in food-mediated intestinal barrier disorders and the resulting symptoms. To analyze the activation of basophils and whether they react to particular food antigens, blood samples are incubated with different staple foods. Basophils carry antigen specific IgE antibodies on their surface. If a cross-reaction with one of the tested food antigens occurs, the cells upregulate the activation marker CD63 on their surface. After stimulation, the samples are stained with antibodies against the general basophil marker CCR3 as well CD63 and the samples are analyzed via flow cytometry to detect basophils positively stained for CCR3 as well as CD63 (activated basophils).
Phenotypic analysis of PBMCs (peripheral blood mononuclear cells) isolated from the blood | week 0, 12, 24
  PBMCs are isolated from blood samples, cultured in cell culture and thereafter, are phenotypically analyzed by fluorescence activated cell sorting (FACS) in order to investigate the influence of nutrition on the immune system.
Analysis of inflammatory markers in the stool (Calprotectin) | week 0, 12, 24
  The concentrations of different inflammatory markers such as Calprotectin are analyzed in the stool to evaluate the intestinal inflammation status quantitatively.
Analysis of fecal biomarkers to evaluate the integrity of the intestinal barrier (Zonulin) | week 0, 12, 24
  The concentrations of fecal biomarkers such as Zonulin are determined to quantitatively evaluate the integrity of the intestinal barrier.
Determination of the I-FABP concentration in the serum | week 0, 12, 24
  The I-FABP concentration is measured in serum samples to evaluate the intestinal permeability. I-FABP is a protein exclusively found in intestinal epithelial cells. If the intestinal epithelium is damaged, I-FABP is released into the circulation and can be measured in the serum. Therefore, I-FABP serum levels are a valid biomarker for intestinal permeability in coeliac disease, wheat sensitivity and also in inflammatory bowel disease.
Determination of the fecal β-Defensin concentration | week 0, 12, 24
  Fecal concentrations of the antimicrobial peptide β-Defensin are determined in the stool.
Fecal microbiome analysis | week 0, 12, 24
  The fecal microbiome is analyzed in stool samples in order to determine the influence and the prebiotic properties of the nutritional therapy (mostly vegetarian Mediterranean wholefood diet) and the additional omission diet on the intestinal microbiome.
Analysis of fecal metabolites | week 0, 12, 24
  Microbial metabolites such as short chain fatty acids (SCFAs) are analyzed in stool samples in order to determine the influence and the prebiotic properties of the nutritional therapy and the additional omission diet on the intestinal microbiome. Prebiotics are nutritional components that promote the growth and activity of beneficial bacterial species. Prebiotics serve as a nutritional basis for these bacteria and promote, for example, their production of SCFAs that act as essential energy substrates for enterocytes and immune cells. These metabolites have been shown to influence immune cell maturation, immune homeostasis, host energy metabolism and the maintenance of mucosal integrity. Therefore, the combined evaluation of microbiome and microbial metabolites in the stool can contribute to a better understanding of the interplay of these factors in the development and treatment of IBD.
Metabolite profiling in the urine | week 0, 12, 24
  Metabolite profiling is done from urine samples. This can also provide valuable insights into the (dys)regulation of gut microbial metabolism and host-microbe co-metabolism in the context of IBD.
Analysis of the composition of bile fluid | week 0, 12, 24
  Oesophagogastroduodenoscopy (OGD) is performed as part of the routine inpatient care to analyze the inflammatory status and the intestinal barrier. During OGD, a sample of bile fluid is collected by simple aspiration from the duodenum in order to assess the secretion and composition of bile acids and their metabolites. Bile acids and their metabolites can have a significant impact on gut health in IBD patients. They have the capacity to modulate inflammation, alter the microbiome and affect the intestinal barrier integrity by regulating the expression of tight junction proteins that control the permeability of the gut wall.
Metabolome analysis of serum samples | week 0, 12, 24
  Metabolome analyses from serum samples are carried out to investigate the influence of diet and intestinal barrier disorders on the disease-associated metabolic profile of Crohn's disease patients. Metabolome analyses enable the visualization of the metabolic product profile of various biological processes. This also enables the evaluation of pathophysiological changes in the metabolism of Crohn's disease patients that has been shown to be significantly different from the metabolome profile of healthy subjects.
Anamnesis | week 0, 12, 24
  Data collected during anamnesis in the course of the routine inpatient stay such as the course of disease or working ability are documented to enable an evaluation of the participants' medical condition and health status.
Concomitant medication | week 0, 12, 24
  Concomitant medication and especially IBD-related therapy of the study participants is documented throughout the study.
Medical history | week 0, 12, 24
  Information on concomitant diseases and the medical history of the study participants is routinely collected and recorded in the course of the inpatient stay as well as throughout the study participation in order to evaluate the participants' medical condition and health status.
Social demographics | week 0, 12, 24
  Social demographic aspects are collected in order to describe the patient collective of the study participants.
Evaluation of the iron status in the blood | week 0, 12, 24
  The iron status is analyzed in the blood to provide indications of IBD-associated complications such as anemia.
Evaluation of the liver status in the blood | week 0, 12, 24
  The liver status is analyzed in blood samples by measuring e.g. ALT, AST, LDH, gamma-GT and alkaline phosphatase in order to provide indications of IBD-associated complications such as liver dysfunction.
Analysis of inflammatory markers in the stool (Lactoferrin) | week 0, 12, 24
  The concentrations of different inflammatory markers such as Lactoferrin are analyzed in the stool to evaluate the intestinal inflammation status quantitatively.
Analysis of inflammatory markers in the stool (EDN) | week 0, 12, 24
  The concentrations of different inflammatory markers such as Eosinophil-derived Neurotoxin (EDN) are analyzed in the stool to evaluate the intestinal inflammation status quantitatively.
Analysis of inflammatory markers in the stool (PMN-Elastase) | week 0, 12, 24
  The concentrations of different inflammatory markers such as PMN-Elastase are analyzed in the stool to evaluate the intestinal inflammation status quantitatively.
Analysis of fecal biomarkers to evaluate the integrity of the intestinal barrier (α-1-Antitrypsin) | week 0, 12, 24
  The concentrations of fecal biomarkers such as α-1-Antitrypsin are determined to quantitatively evaluate the integrity of the intestinal barrier.

CONTACTS AND LOCATIONS:
Overall Officials: Jost Langhorst, Univ. Prof. Dr. med., Principal Investigator — Universität Duisburg-Essen
Locations (1):
- Sozialstiftung Bamberg, Bamberg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No